CLINICAL TRIAL: NCT01432314
Title: A Phase II Trial of Radiation Therapy, Followed by Transarterial Chemoembolization in Patients With Hepatocellular Carcinoma Invading 1st or 2nd Order Branch of Portal Vein
Brief Title: Efficacy of Radiation Therapy and Transarterial Chemoembolization (TACE) to Treat Hepatocellular Carcinoma (HCC)
Acronym: RTANDTACE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Another phase 2 randomized study has been started by other investigators.
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Han Chu Lee, Asan Medical Center, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCLee3915
Record Dates: First submitted 2011-09-07; First posted 2011-09-12 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: patient's survival; tumor response; safety
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment group (Experimental): Child A Hepatocellular carcinoma patients with unilobar portal vein invasion.
  Interventions: Other: Radiation therapy; Other: Transarterial chemoembolization

INTERVENTIONS:
Other: Radiation therapy — A. Started 1 week after entry. B. Equipment: linear accelerator using 6-15 MV photons (external beam equipment). Computerized treatment planning system will be used to determine the radiation fields and 3D dose distribution.
  C. Target volume: include only the portal vein tumor thrombus and 2 cm margin into the contiguous HCC. Respiratory movement will be tracked (4D-CT).
  D. Dose:
  i) Dose for fraction: 3 Gy, at 5 fractions/week ii) Total dose: 45 Gy E. Criteria for stopping RT i) Development of grade 3 or 4 hepatotoxicity or gastrointestinal complications, as defined by CTCAE ver 4.0. Restart of RT should be within 2 weeks after stopping RT.
  Other Names: RT
Other: Transarterial chemoembolization — A. Start at 2 weeks after completion of RT. B. TACE procedure: cisplatin 2 mg/kg infusion with 5-20 mL of lipiodol emulsion through the target artery of HCC. Gelfoam embolization will be used until to no tumor staining on re-angiography.
  C. At an interval of 8 weeks twice, and then every 3 months until contraindications or complete response develop.
  Other Names: TACE

SUMMARY:
In this study, the investigators are to prospectively evaluate patient's survival, tumor response, and safety of RT followed by TACE in Child A patients with unilobar portal vein invasion.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) invading portal vein represents or predisposes to several disastrous clinical conditions. First, obstruction of portal vein per se or accompanying large arterio-portal shunts can cause a rapid deterioration of hepatic function and development of portal hypertension complications. Second, vascular invasion itself is a risk factor for future extrahepatic metastasis. Third, severe complications including hepatic failure may develop after transarterial chemoembolization (TACE) since both hepatic arterial and portal venous blood flows can be interrupted simultaneously. For these reasons, TACE is not routinely recommended in this clinical setting, although there have been some controversies.

Patients with HCC invading portal vein have a dismal prognosis. In an Asian prospective randomized trial evaluating the efficacy of TACE, the median survival of HCC patients with unilobar portal vein invasion was only 2.6 months in control group. Though it was 5.1 months in TACE group, the difference was not significant statistically. Recent two phase III randomized placebo-controlled trials revealed that sorafenib can prolong the patient's survival in the Barcelona Clinic Liver Cancer (BCLC) advanced stage that includes HCC invading portal vein, and thereby the guideline endorsed by the American Association for the Study of Liver Diseases (AASLD) recommended it as a standard therapy for these patients. However, before the advent of sorafenib, many treatment modalities had been used in Asian countries for these patients. Examples are surgical resection, TACE, hepatic arterial infusion chemotherapy, or radiation therapy (RT). Accordingly, guidelines of many Asian countries still adopt these therapies for patients with portal vein invasion, despite there being no solid evidence.

Radiation was traditionally thought to have a limited role in the treatment of HCC. This concept partly resulted from the limited ability to deliver lethal doses using external beam techniques in the past, since the whole-liver tolerance to radiation was reported to be low. However, recent use of three- or four-dimensional conformal radiation therapy (RT) has permitted the delivery of higher doses of radiation to intrahepatic tumors with no increase or even decrease of radiation-induced toxicities. Accordingly, several recent retrospective studies performed in Asia have suggested that RT combined with transarterial chemoinfusion (TACI) or TACE may have a beneficial effect in HCC patients with portal vein invasion. In our retrospective analysis, the median survival in CTP A patients with unilobar portal vein invasion treated with RT and TACE/I was over 22 months, which was obviously longer than the reported median survival in advanced stage patients by BCLC staging system. The median survival was 6 months in patients who were treated only with TACE/I. However, the survival benefit was not obvious in patients with main portal vein invasion.

Despite these encouraging data, radiation-induced hepatotoxicity is still the major obstacle for the widespread use of RT for the treatment of HCC even with the 3D- or 4D-conformal radiation therapy. The reported incidence of hepatotoxicity after RT was up to 15-20%, but about half of the cases were in fact related to hepatitis B virus (HBV) reactivation, which is preventable with preemptive antiviral therapy. Other factors such as the area of RT field or dose may be related to the occurrence of hepatotoxicity. Techniques to deliver radiation beam are also important and tracking of respiratory movement (4D-RT) can minimize complications.

In our center, radiation therapy is mostly focused on the tumor portions invading portal vein to deliver a sufficient radiation dose and to minimize toxicity. With this approach, we control the tumor portions invading portal vein with RT and remnant parenchymal portions of tumors with TACE. Though TACE also carries a risk of hepatic failure in HCC patients with portal vein invasion, our retrospective analysis (submitted data) showed that it can be performed safely in CTP A patients with HCC invading 1st or 2nd order branch of portal vein if the tumor volume is less than 1/2 of total liver volume. Grade 3 or 4 hepatotoxicity developed in 10% of patients. Although there were slight differences in the protocols, several other studies have also reported the effectiveness and safety of this approach.

However, there are still limitations in interpreting pre-existing data. Since most have been retrospective studies, there could be a high probability that treatment-related toxicities were underestimated and an intention-to-treat analysis was not performed. And also, there have been a wide variability in treatment schedule, or evaluating response to treatment and/or treatment-related toxicities among studies.

Therefore, in this study, we are to prospectively evaluate patient's survival, tumor response, and safety of RT followed by TACE in Child A patients with unilobar portal vein invasion.

ELIGIBILITY:
Inclusion Criteria:

* 18 and older than 18 years, and less than 70 years
* Histologically diagnosed HCC, or clinically diagnosed HCC based on the American Association of Study of Liver Disease (AASLD) noninvasive diagnostic criteria for HCC larger than 2 cm in diameter (Patients with chronic HBV or HCV infection, and/or evidence of liver cirrhosis, and typical enhancement pattern (arterial enhancement and portal or delayed washout) on dynamic computed tomography (CT) or magnetic resonance imaging (MRI), or mass with serum alpha fetoprotein level more than 200 ng/mL)
* Treatment naïve HCC patients or patients who received a locoregional therapy(-ies) (radiofrequency ablation, percutaneous ethanol injection, surgical resection; TACE is not allowed) to nontarget lesion at least 3 months prior to baseline scan
* HCC invasion to 1st or 2nd order branch of portal vein
* HCC greater than 2 cm and the tumor volume should be less than half of total liver volume
* CTP score 6 or less than 6 (Child A class only)
* ECOG performance status 0 or 1
* Women with childbearing potential and men must agree to use adequate contraception prior to study entry and during study participation
* Patients who refuse to use sorafenib
* The patient must give written, informed consent

Exclusion Criteria:

* Age of 70 and older, or younger than 18
* HCC less than 2 cm, or tumor volume larger than half of total liver volume
* Invasion to both right and left portal veins, or main portal vein
* Invasion to hepatic vein or inferior vena cava
* Presence of extrahepatic metastasis
* Recurred HCC after liver transplantation
* Prior history of any treatment to target lesion
* Any history of previous RT, TACE, sorafenib or other systemic therapy
* Prior locoregional therapy (radiofrequency ablation, percutaneous ethanol injection therapy, surgery) within 3 months before baseline scan
* CTP score more than 6 (Child class B or C)
* ECOG performance status more than 1
* Presence of ascites or encephalopathy
* Absolute neutrophil count less than 1,000/mm3
* Platelet count less than 60,000/mm3
* INR of prothrombin time more than 1.5
* Serum creatinine more than 1.5 mg/dL
* AST or ALT more than 5x upper limit normal(ULN)(200 IU/L)
* Bilirubin more than 3 mg/dL
* Recent gastrointestinal bleeding including variceal bleeding within 3 months
* History of active gastro-duodenal ulcers within the past 6 months. However, the patient is eligible if a more recent gastroscopy shows complete healing of ulcers.
* Major surgery or serious non-healing wounds within 3 months of start of RT
* Pregnancy or breastfeeding. All female patients with childbearing potential must have a negative pregnancy test within 7 days prior to enrollment.
* Previous or concurrent cancer that is distinct in primary site or histology from HCC, except cervical carcinoma in situ, treated basal cell carcinoma, and superficial bladder tumors (Ta, Tis and T1) (Any cancer curatively treated at least 3 years prior to entry is permitted).
* Any active clinically serious infections (Grade 3, CTCAE version 4.0)
* History of human immunodeficiency virus (HIV) infection
* History of organ allograft
* Patients who agree to use sorafenib

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Time to tumor progression | participants will be followed for the duration of hospital stay and outpatient visit, an expected average of 18 weeks
  At the visiting time of D8, D15, D22, and D29, patients can visit at the outpatient clinic within the window period of ± 1 week. In addition, at the visiting time of D43, D71, D99, and W18, patients can visit at the outpatient clinic within the window period of ± 2 week.
  Progression of target region or appearance of new lesion will be checked at every visit.

SECONDARY OUTCOMES:
Progression-free survival of HCC patients | participants will be followed for the duration of hospital stay and outpatient visit, an expected average of 18 weeks
  At the visiting time of D8, D15, D22, and D29, patients can visit at the outpatient clinic within the window period of ± 1 week. In addition, at the visiting time of D43, D71, D99, and W18, patients can visit at the outpatient clinic within the window period of ± 2 week.
safety of RT followed by TACE | participants will be followed for the duration of hospital stay and outpatient visit, an expected average of 18 weeks
  At the visiting time of D8, D15, D22, and D29, patients can visit at the outpatient clinic within the window period of ± 1 week. In addition, at the visiting time of D43, D71, D99, and W18, patients can visit at the outpatient clinic within the window period of ± 2 week.
  Safety evaluation will be performed according to the Common Terminology Criteria for Adverse Events (CTCAE; version 4.0).
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability
Overall survival of HCC patients | participants will be followed for the duration of hospital stay and outpatient visit, an expected average of 18 weeks
  At the visiting time of D8, D15, D22, and D29, patients can visit at the outpatient clinic within the window period of ± 1 week. In addition, at the visiting time of D43, D71, D99, and W18, patients can visit at the outpatient clinic within the window period of ± 2 week.
Time to TACE discontinuation | participants will be followed for the duration of hospital stay and outpatient visit, an expected average of 18 weeks
  At the visiting time of D8, D15, D22, and D29, patients can visit at the outpatient clinic within the window period of ± 1 week. In addition, at the visiting time of D43, D71, D99, and W18, patients can visit at the outpatient clinic within the window period of ± 2 week.
Best tumor response by modified RECIST (mRECIST) and RECIST criteria | participants will be followed for the duration of hospital stay and outpatient visit, an expected average of 18 weeks
  At the visiting time of D8, D15, D22, and D29, patients can visit at the outpatient clinic within the window period of ± 1 week. In addition, at the visiting time of D43, D71, D99, and W18, patients can visit at the outpatient clinic within the window period of ± 2 week.

CONTACTS AND LOCATIONS:
Overall Officials: Han Chu Lee, M.D, Principal Investigator — Department of Internal Medicine, Asan Liver Center, Asan Medical Center, University of Ulsan College of Medicine